CLINICAL TRIAL: NCT05540587
Title: A Randomized, Open, Phase 2 Study to Evaluate the Efficacy and Safety of Edoxaban in Patients With Atrial Fibrillation and Mitral Stenosis
Brief Title: Efficacy and Safety of Edoxaban in Patients With Atrial Fibrillation and Mitral Stenosis
Acronym: ERTEMIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sung-Hwan Kim (Other)
Collaborators: Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Sung-Hwan Kim, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC21MIDS0296
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Mitral Valve Stenosis; Atrial Fibrillation; Stroke; Systemic Embolism
Keywords: Edoxaban; Warfarin; Stroke; Systemic embolism; Mitral Valve Stenosis; Atrial Fibrillation
MeSH Terms: conditions — Mitral Valve Stenosis; Atrial Fibrillation; Stroke | interventions — edoxaban; Warfarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban (Experimental): Patients in the Edoxaban group take Edoxaban 60mg once daily. If any of the following conditions are present, take 30mg once daily.
  * CrCl 15-50mL/min
  * Body weight ≤ 60kg
  * Concomitant use of P-glycoprotein inhibitor (Dronearone, Ciclosporine, Erythromycin or Ketoconazole)
  Interventions: Drug: Edoxaban
- Warfarin (Active Comparator): Patients in the Warfarin group take Warfarin 2-10mg once daily, dose adjusted with the target INR 2-3. In the elderly or frail patients, a lower dose administration is allowed at the discretion of the investigator.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Edoxaban — Patients in the Edoxaban group take Edoxaban 60mg once daily. If any of the following conditions are present, take 30mg once daily.
  * CrCl 15-50mL/min
  * Body weight ≤ 60kg
  * Concomitant use of P-glycoprotein inhibitor (Dronearone, Ciclosporine, Erythromycin or Ketoconazole)
  Arms: Edoxaban
Drug: Warfarin — Patients in the Warfarin group take Warfarin 2-10mg once daily, dose adjusted with the target INR 2-3. In the elderly or frail patients, a lower dose administration is allowed at the discretion of the investigator.
  Arms: Warfarin

SUMMARY:
This study aims to compare the efficacy and safety of the edoxaban and the warfarin in atrial fibrillation patients with mitral stenosis.

The study design is a multicenter, randomized, open-label, investigator initiated phase 2 trial. The patients were randomly assigned to Edoxaban or Warfarin groups. Primary outcome was a composite of stroke and systemic arterial thromboembolism. The safety outcome was major bleeding.

DETAILED DESCRIPTION:
Non-vitamin K antagonist oral anticoagulants (NOACs) are generally recommended as 1st line therapy for oral anticoagulant in patients with atrial fibrillation (AF). But, the efficacy and safety of NOAC in AF patients with prosthetic mechanical heart valves or moderate to severe mitral valve stenosis have not been proven, and the guidelines recommend vitamin K antagonist (VKA) administration to those patient groups. This trial aims to compare the efficacy and safety of the edoxaban and the warfarin in AF patients with moderate to severe mitral valve stenosis.

Edoxaban in patients with aTrial fibrillation and MItral Stenosis (ERTEMIS) trial is a multicenter, randomized, open-label, investigator initiated phase 2 trial. The patients were randomly assigned to Edoxaban or Warfarin groups. The primary efficacy outcome is a composite of stroke and systemic arterial thromboembolism. The secondary efficacy outcomes are each component of the primary efficacy outcomes and death from any cause. The safety outcome was major bleeding.

ELIGIBILITY:
* Inclusion criteria

  * 18 < Age < 80
  * AF diagnosed by ECG at any time prior to enrollment
  * Moderate or severe mitral valve stenosis diagnosed by echocardiography at any time prior to enrollment
* Exclusion criteria

  * Refusal to consent
  * Transient AF due to reversible cause (Postoperative, ongoing systemic inflammation, thyrotoxicosis)
  * Patients undergoing mechanical valve replacement
  * Coagulopathy
  * Hepatic impairment with significant bleeding risk
  * High bleeding risk due to following disease or condition diagnosed within 1 month prior to randomization

    * GI ulcer or bleeding, Esophageal or gastric varix, Malignancy, Brain or cord injury, Surgery for brain, spinal cord, opthalmic, Intracranial hemorrhage, Arteriovenous malformation, Vascular aneurysms, Brain or spinal vascular disorder
  * Stroke, Systemic arterial thromboembolism, Acute myocardial infarction diagnosed within 14 days prior to randomization
  * End stage kidney disease (CrCL < 15mL/min) or Dialysis
  * Severe hypertension
  * Alcohol abuse or other psychiatric disease
  * Epidural puncture or anesthesia
  * Pulmonary thromboembolism with hemodynamical instability requiring thrombolysis or thrombectomy
  * Pregnant or lactating women
  * Allergy to edoxaban or warfarin
  * Ongoing need for other anticoagulant or clarithromycin, rifampin)
  * Participants for other trials within 1 month prior to enrollment
  * Other patients to be inappropriate to participate in the trial determined by the investigator

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Composite of Stroke or Systemic arterial thromboembolism | 15 days after randomization
  The number of patients with the first occurrence of a stroke or systemic embolism during the study period

SECONDARY OUTCOMES:
Stroke | 15 days after randomization
  The number of patients with the first occurrence of a stroke during the study period
Systemic embolism | 15 days after randomization
  The number of patients with the first occurrence of a systemic embolism during the study period
Death from any cause | 15 days after randomization
  The number of patients who died for any reason during the study period

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Seoul St. Mary's Hospital, Seoul, Seocho-gu
  - Yeouido St. Mary's hospital, Yeongdeungpo-gu, Seoul
  - Bucheon St. Mary's hospital, Bucheon-si
  - Daejeon St. Mary's hospital, Daejeon
  - Incheon St. Mary's hospital, Incheon
  - St. Vincent hospital, Suwon
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si